CLINICAL TRIAL: NCT03545152
Title: Non-pharmacological Interventions on Cognitive Functions in Older People With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu-Ting Huang (Other)
Responsible Party: Sponsor-Investigator, Tzu-Ting Huang, Professor, School of Nursing, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 103-7443B
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Mild Cognitive Impairment; TTM; Physical Activity; Cognitive Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- comparison group (No Intervention): No procedure conducted between the pre- and the post-test evaluations, and they received an abridged version of the training after the post-test session.
- exercise group (Experimental): The exercise program will include instructions on how to read the program, complete the activities, record their sessions, and exercise safely at first day. To promote incorporating exercising in their daily life routine during the 24-week period, we provided 2 group-based (5-8 participants with 2 instructors at community centers, 60' each) and one home-based (with the exercise program VCD and manual to bring home, 30') exercise program.
  Interventions: Behavioral: Exercise; Behavioral: New life-style
- cognitive training group (Experimental): Consisted of 12 weekly sessions, lasting 60-90 minutes in groups of 5-8 participants, and 3 monthly boost sessions (to review the strategies and practice solving problems as well). The main strategy was to use cognitive rehabilitation strategies to promote generalization in this process to improve memory and behavior.
  Interventions: Behavioral: Cognitive training; Behavioral: New life-style

INTERVENTIONS:
Behavioral: Exercise — Prescription exercise: frequency, intensity, type, time, and progression (FITT-PRO).
  150 min/week (the intensity will be moderate). exercise routine: warming up, resistance training and aerobic exercise training(range of motion and flexibility exercises)
  Arms: exercise group
Behavioral: Cognitive training — Cognitive training intervention consisted of 12 weekly sessions, lasting 60-90 minutes in groups of 5-8 participants, and 3 monthly boost sessions (to review the strategies and practice solving problems as well). The main strategy was to use cognitive rehabilitation strategies to promote generalization in this process to improve memory and behavior.
  Arms: cognitive training group
Behavioral: New life-style — Combination of exercise and cognitive interventions
  Arms: cognitive training group; exercise group

SUMMARY:
This project is proposed to be a three-year project. The purposes of this project are to develop and examine physical activity program, cognitive rehabilitation training, and new life-style (combination of exercise and cognitive) interventions on primary outcomes (cognitive function), and secondary outcomes (physical fitness, QOL and depression) among community-dwelling elderly adults with MCI.

DETAILED DESCRIPTION:
Aim. develop and examine physical activity program, cognitive rehabilitation training, and new life-style (combination of exercise and cognitive) interventions on primary outcomes (cognitive function), and secondary outcomes (physical fitness, QOL and depression) among community-dwelling elderly adults with MCI.

Background. Mild cognitive impairment (MCI) is a common clinical syndrome that identifies people at high risk of developing dementia, and the prevalence range from 7.7 to 51.7%. Although treatments for MCI are currently unavailable, preliminary evidence has identified potential neuro-protective effects of exercise program and cognitive rehabilitation, which may lead to improved outcomes. However, the design and delivery of an appropriate program for people with MCI is challenging for having physical, psychological, cognitive, and social barriers.

Design. A prospective randomized control trial. We developed a Physical activity stage-matched intervention (SMI) (1st year), cognitive rehabilitation (2nd year) and New lifestyle program

ELIGIBILITY:
Inclusion Criteria:

* had a subjective memory complaint
* MMSE score<16, 21 or 24, based on their years of education (illiterate, 6 or >9 years, respectively, Yeh et al., 2000), but needed >13 or objective memory impairment: AQ>5 or at least one item of IADL dependence
* able to carry out activities in daily life

Exclusion Criteria:

* using walking devices
* depression or dementia diagnosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 192 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination | 8min
  The participants' cognitive function was assessed by the Mini-Mental State Examination (cut point base for participants' levels of education).
The Alzheimer's Questionnaire | 2min
  Malek-Ahmadi et al., (2012) a 21-item, informant-based dementia assessment designed for ease of use in a primary care setting.
Taiwan version of Prospectiv and Retrospective Memory Questionaire (PRMQ) | 5min
  There are 11 items and include general memory and prospective memory sections for analysis the type and frequency of memory problem in elders' daily live. Items are posed in likert scale ranges from 1 (never) to 5 (always). The total score may range from 11-55. A higher score indicates a higher level of memory impaired.

SECONDARY OUTCOMES:
Mobility | 10min
  The Tinetti Performance-Oriented Mobility Assessment (POMA) is a balance tool that was originally developed for use in the institutionalized, older adult population and contains both a balance and a gait component (Tinetti, 1986). The test comprises 16 items (9 balance-related items and 7 gait-related items), with the highest achievable score being 28 points
Depressive symptoms | 3min
  A short-form Geriatric Depression Scale (GDS) that consisted of 15 questions was the primary outcome measure (Sheikh and Yesavage, 1986). Scores of 0-4 are considered normal; 5-8 indicates mild depression; 9-11 indicates moderate depression; and 12-15 indicates severe depression. The Chinese version of the GDS-15 demonstrates high reliability (Liao et al., 2005); in this study, the Cronbach's α is .91.
Quality of life | 8min
  The SF-36 questionnaire was used to measure quality of life. This 36-item questionnaire assesses health-related functions for eight distinct domains, which can be divided into physical component and mental component scales. Subsequent to summing the Likert-scaled items in the SF-36 survey, scores in each scale are standardized so that they each range from 0 to 100.